CLINICAL TRIAL: NCT04058379
Title: Artificial Intelligence Analysis of Initial Scan Evolution of Traumatic Brain Injured Patient to Predict Neurological Outcome: Pilot Translational an Exploratory Study
Brief Title: Artificial Intelligence Analysis of Initial Scan Evolution of Traumatic Brain Injured Patient to Predict Neurological Outcome
Acronym: RADIOMIC-TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38RC19.193
Record Dates: First submitted 2019-07-15; First posted 2019-08-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-11

CONDITIONS: Trauma, Brain
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT scan (Experimental): During this study each patient will have 3 CT scans : D0, D1 and D3. A daily follow up during first seven days in ICU, then a follow up at D28 if still in hospital, and a phone call at M6 for neurological outcome
  Interventions: Radiation: CT scan

INTERVENTIONS:
Radiation: CT scan — 3 ct scans : D0, D1 and D3

SUMMARY:
We assume that an early iterative automatic CT scan analysis (D0, D1 and D3) by different AI approaches will allow an early differentiation of the tissues evolution after TBI. Our objective is to couple theses scan profiles to a neurological evolution, measured by therapeutic intensity.

DETAILED DESCRIPTION:
Traumatic brain injury is a common and serious pathology, responsible of an important morbi-mortality. The TBI can be consider as a complex set of nosological entities of different evolution with difficult early identification whereas the main issue of this pathology depends on prevention and management of the lesions caused by the initial cerebral aggression.

Different evolutionary profiles seems to exist and sometimes coexists: edema evolution, hemorrhagic transformation and/or cerebrospinal fluid (CSF) resorption issues with hydrocephalus apparition.

Currently, there is no Imaging methods that can be used in every day clinical management that allows a visualization, quantification and prediction of these different lesional evolutions

CT scan is the reference imaging method for TBI patient monitoring. It allows a lesion description, a therapeutic adaptation and an evaluation of the prognostic.

Even if it is used as a routine examination, the analysis of cerebral scanners remains manual and a non-quantitative one, which make a little informative analysis as far as lesions evolution is concerned.

Recently it has been established the automatic MRI analysis with AI approach allows:

1. - To show aspects of images that can't be seen to the naked eye
2. - To automatically segment and quantify the different tissues (edema, hemorrhage...). First tests on this kind of analysis on CT scans shows that this technology can be transferred from MRI to CT scans and more importantly it brings out new quantitative informations on cerebral lesions evolution.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Closed TBI
* Primary admission in Grenoble University Hospital
* Initial CT scan with visible cerebral lesion rated at least 3 on abbreviated injury score (AIS)
* In ICU for an expected length of 48 hours
* Social security system affiliation

Exclusion Criteria:

* Life expectation <48 hours
* In ICU for more than 24h
* Transferred from another hospital
* Patients corresponding to articles L1121-5, L1121-6, L1121-7, L1121-8 (under legal protection) of French Public Health Code
* Patient in exclusion time of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-10-12 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution during first 7 days in ICU with therapeutic intensity level (TILsum) | 7 days after TBI
  Composite criteria : Head position, depth, sort and objective of sedation, presence or absence of a CSF draining system, management of ventilation, presence or absence of a hyperosmolar therapy, management of body temperature, surgical intervention for intracranial hypertension.

SECONDARY OUTCOMES:
Mortality according to scan profiles | 28 days after TBI and 6 month after TBI
Morbidity (consequences of the trauma) according to scan profiles | 28 days after TBI
  Lenght of stay in ICU with more than 20 mmHg of intracranial pressure with no stimulation
Morbidity (consequences of the trauma) according to scan profiles | 28 days after TBI
  length of stay in ICU with a therapeutic intensity level > or = 8,
Morbidity (consequences of the trauma) according to scan profiles | 28 days after TBI
  Hospital stay length
Morbidity (consequences of the trauma) according to scan profiles | 28 days after TBI
  ICU stay length days with mechanical ventilation
Morbidity (consequences of the trauma) according to scan profiles | 6 months after TBI
  Glasgow Outcome Scale (GOSe)
Comparison and Description of correlation between early scan profiles evolution signature by AI and to clinical evolution (with TILSum) | 7 days after TBI
  Analysis of main outcome (TIL sum after 7 days in ICU maximum) according to a kinetic scan evolution between D0, D1 and D3
Neurological Pupil Index | 1 day after TBI
  Measure of neurological pupilla index within 1h after admission and at D1

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOUZAT, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brossard C, Greze J, de Busschere JA, Attye A, Richard M, Tornior FD, Acquitter C, Payen JF, Barbier EL, Bouzat P, Lemasson B. Prediction of therapeutic intensity level from automatic multiclass segmentation of traumatic brain injury lesions on CT-scans. Sci Rep. 2023 Nov 17;13(1):20155. doi: 10.1038/s41598-023-46945-9. PMID 37978266